CLINICAL TRIAL: NCT02372396
Title: A Proof of Concept and Feasibility Trial of Compassion Meditation for PTSD
Brief Title: Compassion Meditation for PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Veterans Medical Research Foundation (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Ariel Lang, PhD, Research Psychologist, Veterans Medical Research Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H130565; 1R34AT007936-01A1 (NIH)
Record Dates: First submitted 2015-02-03; First posted 2015-02-26 (Estimated); Results first posted 2018-09-05 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; Psychotherapy; Operation Enduring Freedom/Operation Iraqi Freedom (OEF/OIF); Veterans
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Compassion Meditation (Experimental): Compassion Meditation delivered in 10 2-hour group treatment sessions.
  Interventions: Behavioral: Compassion Meditation (CM)
- Relaxation (Active Comparator): Relaxation delivered in 10 2-hour group treatment sessions.
  Interventions: Behavioral: Relaxation

INTERVENTIONS:
Behavioral: Compassion Meditation (CM) — Compassion meditation is a meditative practice focused on the wish that others and the self may be free of suffering. Because this particular form of meditation has been shown to elicit positive emotion and feelings of connection with other people, it is uniquely well suited to addressing PTSD, which is characterized by strong negative affect, deficits in positive emotion and social connectedness.
  Other Names: CM
  Arms: Compassion Meditation
Behavioral: Relaxation — Relaxation Training is selected as the control condition because it is a good match for nonspecific aspects of the meditative practice (e.g., attention, support, contact with a mental health provider) and it is structurally similar to meditation (e.g., restful, in session and at home exercises).
  Arms: Relaxation

SUMMARY:
The goal of this project is to refine an existing compassion meditation protocol for individuals with posttraumatic stress disorder (PTSD), to examine the safety and feasibility of this approach and to collect data to make initial estimates of efficacy.

DETAILED DESCRIPTION:
There is considerable public and professional interest in complementary and alternative approaches, including meditation, for managing posttraumatic stress disorder (PTSD), but there is little empirical support to guide their use. Multiple meditative techniques can be applied to the amelioration of this disorder, and the literature suggests that they operate by different mechanisms. Compassion meditation is a meditative practice focused on the wish that others and the self may be free of suffering. Because this particular form of meditation has been shown to elicit positive emotion and feelings of connection with other people, it is uniquely well suited to addressing PTSD, which is characterized by strong negative affect, deficits in positive emotion and social connectedness.

Compassion meditation has not been evaluated for use with PTSD patients; therefore, the goal of this project is to refine an existing compassion meditation protocol for individuals with PTSD, to examine the safety and feasibility of this approach and to collect data to make initial estimates of efficacy. The proposed project will be completed in two phases.

In phase one, the compassion meditation protocol will be executed with individuals with PTSD and iteratively refined based on therapist and participant feedback. In addition, a relaxation protocol that was used in a previous PTSD trial will be modified to match the length and format of the meditative practice.

In phase two, the investigators will complete a pilot study to examine the feasibility of conducting a randomized trial comparing these interventions and to provide information that will allow us to better design future projects. Ultimately, the research informed by this project may provide an additional option for treatment of PTSD, which would be an important contribution because existing treatment approaches are not universally acceptable or effective.

ELIGIBILITY:
Inclusion Criteria:

* Veteran of at least 18 years of age
* PTSD as defined by the Diagnostic and Statistical Manual Version 5 (DSM-5)
* Capacity to consent
* Willing to commit to 8 consecutive weekly sessions lasting 2 hours in duration and to complete assessment materials.

Exclusion Criteria:

* Serious suicidality or homicidality that has required urgent or emergent evaluation or treatment within the past three months
* A known, untreated substance use disorder (inclusion is possible if there is evidence that the individual has been afforded and is complying with treatment for the substance problem)
* Serious Axis I mental disorders, such as psychotic disorders or bipolar type I, or serious dissociative symptoms
* Cognitive impairment that would interfere with consent or treatment
* Circumstances that lead to recurrent traumatization (e.g., engaged in a violent relationship)
* Concurrent enrollment in any other treatment specifically targeting PTSD symptoms or social functioning (e.g., couples therapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ariel J Lang, PhD, Principal Investigator — San Diego Veterans Healthcare System
Locations (1):
- VA San Diego Healthcare System, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- CBCT-Vet: Cognitively Based Compassion Training, Veteran Version (CBCT-Vet) delivered in 10 1.5-hour group treatment sessions.
  CBCT-Vet is a compassion meditation practice focused on the wish that others and the self may be free of suffering. Because this particular form of meditation has been shown to elicit positive emotion and feelings of connection with other people, it is uniquely well suited to addressing PTSD, which is characterized by strong negative affect, deficits in positive emotion and social connectedness.
- Veteran.Calm: Veteran.calm delivered in 10 1.5-hour group treatment sessions.
  Veteran.calm is a form of relaxation training that was selected as the control condition because it is a good match for nonspecific aspects of the meditative practice (e.g., attention, support, contact with a mental health provider) and it is structurally similar to meditation (e.g., restful, mind-body focus, in session and at home exercises).
Period: Overall Study
Arm/Group | CBCT-Vet | Veteran.Calm
Started | 17 | 20
Began Intervention | 14 | 14
Completed | 10 | 11
Not Completed | 7 | 9
Not completed — Lost to Follow-up | 7 | 9

BASELINE CHARACTERISTICS:
Groups:
- CBCT-Vet: CBCT-Vet delivered in 10 1.5-hour group treatment sessions.
  CBCT-Vet is a compassion meditation practice focused on the wish that others and the self may be free of suffering. Because this particular form of meditation has been shown to elicit positive emotion and feelings of connection with other people, it is uniquely well suited to addressing PTSD, which is characterized by strong negative affect, deficits in positive emotion and social connectedness.
- Total: Total of all reporting groups
Arm/Group | CBCT-Vet | Veteran.Calm | Total
Number analyzed (Participants) | 17 | 20 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data presented on participants who began the intervention rather than on the intent-to-treat sample.
  years
    number analyzed (Participants) | 14 | 14 | 28
    (all) | 45.5 (16.6) | 52.7 (11.4) | 49.11 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Presenting data on those who began treatment
  Participants
    number analyzed (Participants) | 14 | 14 | 28
    Female | 4 | 3 | 7
    Male | 10 | 11 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Presenting data on those who initiated treatment
  Participants
    number analyzed (Participants) | 14 | 14 | 28
    Hispanic or Latino | 2 | 8 | 10
    Not Hispanic or Latino | 12 | 6 | 18
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Presenting data on those who began treatment
  Participants
    number analyzed (Participants) | 14 | 14 | 28
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 1 | 1 | 2
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    Black or African American | 5 | 1 | 6
    White | 7 | 7 | 14
    More than one race | 0 | 5 | 5
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 20 | 37

OUTCOME MEASURES:

1. Primary Outcome: Clinician Administered PTSD Scale -5 (CAPS-5) PTSD Severity
Description: Clinical interview that quantifies PTSD symptomatology according to DSM-5, generating a continuous measure of severity (range 0-80) where higher scores indicate more symptomatology
Time Frame: Baseline and 10 weeks
Population: Completer analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBCT-Vet | Veteran.Calm
Number analyzed (Participants) | 10 | 11
units on a scale
  Baseline | 35.8 (13.9) | 37.9 (11.9)
  10 weeks | 20.4 (11.8) | 35.3 (7.7)

ADVERSE EVENTS:
Time Frame: 12 weeks (duration of participant involvement)
Arm/Group | CBCT-Vet | Veteran.Calm
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/20
Other Adverse Events (participants affected / at risk) | 0/17 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-09-15): https://cdn.clinicaltrials.gov/large-docs/96/NCT02372396/Prot_SAP_000.pdf